CLINICAL TRIAL: NCT01064986
Title: The Effects of Hydrocortisone in Endotoxemia in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 0220070126; NIH/DHHS (Other Grant/Funding Number: GM34695)
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Infections
Keywords: Immune System
MeSH Terms: conditions — Infections | interventions — Endotoxins; Lipopolysaccharides; Sodium Chloride; Epinephrine; hydrocortisone hemisuccinate; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): IV Endotoxin plus saline vehicle (placebo)
  Interventions: Biological: Endotoxin, Lipopolysaccharide, LPS; Biological: Placebo
- B (Active Comparator): IV Endotoxin plus IV hydrocortisone
  Interventions: Biological: Endotoxin, Lipopolysaccharide, LPS /Epinephrine; Biological: Hydrocortisone

INTERVENTIONS:
Biological: Endotoxin, Lipopolysaccharide, LPS — Clinical Center Reference Endotoxin, lot 2, sterile saline, 1 ng/kg, bolus IV administration (~5 minutes)
  Other Names: Sodium Chloride Solution
  Arms: A
Biological: Endotoxin, Lipopolysaccharide, LPS /Epinephrine — Clinical Center Reference Endotoxin, lot 2, sterile saline, 1 ng/kg, continuous IV administration (Hydrocortisone 3mcg/kg/min)
  Other Names: Solu-Cortef
  Arms: B
Biological: Placebo — Saline vehicle (placebo)
  Arms: A
Biological: Hydrocortisone — Hydrocortisone
  Arms: B

SUMMARY:
Corticosteroids are substances produced by the adrenal gland to help the body fight against infection or injury. Hydrocortisone is a man-made form of this substance. Endotoxin is a man-made substance, which causes the body to "mimic" sickness(fever,chills,and achiness)for a few hours. This study is designed to give hydrocortisone before and after Endotoxin to determine if this medication can prevent or relieve any of the symptoms caused by the Endotoxin.

DETAILED DESCRIPTION:
The body's immune response to injury otr infection is very complex. Immune cell activity, the release of specific mediators (such as proteins), genetics (Deoxyribonucleic acid or DNA) and/or the body's "instructions" for making proteins (Ribonucleic Acid or RNA) may effect the body's clinical response to a stress such as an infection.Hydrocortisone is a substance produced by the body (in the adrenal gland)in response to stress such as infection or injury. Endotoxin is a man- made substance, which causes the body to "mimic" sickness (fever, chills, and achiness) for a few hours. This study is designed to give hydrocortisone before and/or after endotoxin to determine if this medication can prevent or relieve any of the symptoms caused by endotoxin.In addition, this study may determine whether any of the above(proteins,DNA,RNA,etc.) correlate with or affect the body's response to hydrocortisone and/or endotoxin. This will enable the investigator to better understand whether treatment with this substance can alter the body's immune response.

ELIGIBILITY:
Inclusion Criteria:

* General good health as demonstrated by medical history, physical& laboratory tests
* Age between 18 and 40 years
* Written informed consent prior to the performance of any study related procedures

Exclusion Criteria:

* History of cancer, rheumatoid arthritis, or immunological, renal, hepatic, endocrine, neurologic, heart disease or hypertension
* Any medication taken in past 48 hrs (except birth control)
* Recent history of alcohol or drug abuse
* Unable to provide written informed consent
* Exposure to any experimental agent or procedure within 30 days of study
* Pregnant or breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Physiological, Hematological, Immunological Responses | 0.5-24 hrs post Endotoxin administration

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Corbett, MD, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Rutgers-RWJMS, New Brunswick, New Jersey, United States